CLINICAL TRIAL: NCT01200940
Title: Metabolic Effects of Non-Nutritive Sweeteners
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 100163; 10-DK-0163
Record Dates: First submitted 2010-09-11; First posted 2010-09-14 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: GLP-1; Glucose Tolerance; Gut Hormones
MeSH Terms: interventions — trichlorosucrose; Aspartame; acetosulfame

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Phase I - Low-dose sweetener (Experimental): 68 mg sucralose dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Sucralose
- Phase I - Medium-dose sweetener (Experimental): 170 mg sucralose dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Sucralose
- Phase I Control Condition (Placebo Comparator): 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Control
- Phase I- High-dose sweetener (Experimental): 250 mg sucralose dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test.
  Interventions: Other: Sucralose
- Phase II - Control Condition (Placebo Comparator): 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Control
- Phase II - Diet Soda 1 (Experimental): less than or equal to 5mg/kg sucralose, less than or equal to 15 mg/kg acesulfame-potassium dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Sucralose; Other: Acesulfame-Potassium
- Phase II - Diet Soda 2 (Experimental): less than or equal to 5 mg/kg sucralose, less than or equal to 50 mg/kg aspartame, less than or equal to 15 mg/kg acesulfame-potassium dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Sucralose; Other: Aspartame; Other: Acesulfame-Potassium
- Phase II - Water with sucralose and acesulfame-potassium (Experimental): less than or equal to 5mg/kg sucralose, less than or equal to 15 mg/kg acesulfame-potassium dissolved in 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Interventions: Other: Sucralose; Other: Acesulfame-Potassium

INTERVENTIONS:
Other: Sucralose — sucralose will be given at doses of 68 mg (equivalent to one 12 oz soda) 170 mg (equivalent to two and one-half 12 oz sodas, and 250 mg (equal to 100% of the FDA s acceptable daily intake for a 50kg individual).
  Arms: Phase I - Low-dose sweetener; Phase I - Medium-dose sweetener; Phase I- High-dose sweetener; Phase II - Diet Soda 1; Phase II - Diet Soda 2; Phase II - Water with sucralose and acesulfame-potassium
Other: Aspartame — To determine the impact of sucralose and acesulfame- potassium ( aspartame) together on GLP-1 secretion, satiety, and the rate of intestinal glucose absorption. The doses of sucralose and acesulfame- potassium reflect the sweetener concentrations in the previously used Diet Rite Cola .
  Arms: Phase II - Diet Soda 2
Other: Acesulfame-Potassium — To determine the impact of sucralose and acesulfame- potassium ( aspartame) together on GLP-1 secretion, satiety, and the rate of intestinal glucose absorption. The doses of sucralose and acesulfame- potassium reflect the sweetener concentrations in the previously used Diet Rite Cola .
  Arms: Phase II - Diet Soda 1; Phase II - Diet Soda 2; Phase II - Water with sucralose and acesulfame-potassium
Other: Control — 360 mL of water will be drunk 10 minutes prior to a 75 g oral glucose tolerance test
  Arms: Phase I Control Condition; Phase II - Control Condition

SUMMARY:
Background:

- Artificial sweeteners, such as sucralose (brand name Splenda), are very commonly found in products such as diet soft drinks. Recently, researchers learned that these sweeteners may affect hormones in the body, especially when they are consumed in combination with real sugar. Changes in hormone levels may, in turn, result in changes in blood sugar, appetite, and weight. Researchers are interested in studying the effects of artificial sweeteners on the metabolism and hormonal levels of healthy volunteers.

Objectives:

* To study the effects that artificial sweeteners have on hormone levels, blood sugar, and appetite.
* To evaluate whether artificial sweeteners change the rate at which food passes out of the stomach into the gut, or the rate at which the body absorbs sugar from the gut.
* To evaluate the effects that different amounts of artificial sweeteners have on hormone levels.

Eligibility:

- Healthy volunteers between 18 and 45 years of age.

Design:

* This study will require one screening visit and four testing visits, scheduled on different days.
* At the screening visit, eligible participants will be screened with a physical examination, medical history, blood samples, and body measurements (including height, weight, body circumferences, and skin folds). Participants will also be asked about how much artificial sweetener they typically consume and will have taste tests, in which a small amount of flavored liquid is placed on the tongue and participants will name the flavor and rate its intensity.
* Participants will have four glucose tolerance tests on four different days. In preparation for the test, participants will not eat or drink anything but water for 12 hours prior to the test. Blood will be drawn before the test, and participants will drink one of the following study liquids, selected at random:
* Plain water
* Water mixed with sucralose (the amount found in one 12 oz diet soft drink)
* Water mixed with sucralose (the amount found in 2.5 12 oz diet soft drinks)
* Water mixed with sucralose (the amount found in 3.7 12 oz diet soft drinks)
* Ten minutes after drinking the study liquid, participants will have a sugary drink that will allow researchers to measure sugar absorption and the speed with which food leaves the stomach.
* In addition, participants will complete questionnaires about hunger levels before drinking the sugar solution and at regular intervals for 2 hours afterward. Blood samples will be taken at regular intervals as well.

DETAILED DESCRIPTION:
Background

Consumption of non-nutritive sweeteners is common practice in the US, and these chemicals are generally thought to be metabolically inert. However, recent data obtained from animal studies demonstrate that non-nutritive sweeteners play an active metabolic role within the gastrointestinal tract. Sweet-taste receptors, including the T1R family and Alpha-gustducin, respond not only to caloric sugars such as sucrose, but also to non-nutritive sweeteners, including sucralose (Splenda ) and acesulfame-K . In both humans and animals, these receptors have been shown to be present in glucagon-like-peptide-1 (GLP-1) secreting L cells of the gut mucosa as well as in lingual taste buds , and serve as critical mediators of GLP-1 secretion . We have demonstrated in a previous study that diet soda augments glucose-stimulated GLP-1 secretion . In addition, there is evidence in animals that activation of intestinal sweet-taste receptors by non-nutritive sweeteners enhances intestinal glucose absorption via upregulation of the glucose transporter, GLUT2 .

Aims

The purpose of this study is to broadly explore the effects of non-nutritive sweeteners on glucose and glucoregulatory hormones in healthy humans. To this end, we plan the following:

Primary Aim: To confirm that the non-nutritive sweetener sucralose (versus other ingredients in diet soda) augments glucose-stimulated GLP-1 secretion

Secondary Aims:

1. To study whether increased GLP-1 secretion due to non-nutritive sweeteners alters gastric emptying or satiety
2. To determine a dose-response relationship for non-nutritive sweeteners on glucose-stimulated GLP-1 secretion
3. To determine whether non-nutritive sweeteners alter the rate of intestinal glucose absorption
4. To test whether non-nutritive sweeteners affect levels of other incretin or gut hormones

Methods

Healthy men and women ages greater than or equal to 18 years, and prepubertal children ages 6-12 years, across a wide range of body mass indices will participate in a variety of paired experiments, in randomized order, with each subject serving as his or her own control. In each experiment, the subject will ingest either a non-nutritive sweetener or control, and a glucose load (oral glucose tolerance test). The following measurements will be obtained:

1. Serial measurement of glucose, insulin, C-peptide, GLP-1, and other incretin and gut hormones
2. Rate of gastric emptying using acetaminophen labeling in the oral glucose or mixed meal
3. Measurement of hunger and satiety using validated questionnaires
4. Measurement of intestinal glucose absorption using a glucose analog

ELIGIBILITY:
* MAIN STUDY:

INCLUSION CRITERIA:

* Age greater than or equal to 18 years
* No known active medical conditions

EXCLUSION CRITERIA:

* Current use of prescription or non-prescription medication. Certain exceptions are permitted, including topical medications, vitamins, and hormonal contraceptives. Other medications may be permitted at the discretion of the investigators.
* Recent (past 2 months) use of drugs that alter glucose metabolism (e.g. metformin), alter gastric pH (e.g. proton pump inhibitors) or gastric emptying (e.g. metoclopramide)
* ALT or AST more than 1.5 times the upper limit of normal
* Positive urine pregnancy test
* Known allergy, sensitivity or other contraindication to any study food or drug or its vehicle
* Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to provide informed consent, or to comply with study procedures
* Body weight less than 50 kg
* Diabetes (fasting blood glucose of 126 mg/dl or higher, or 2-hour blood glucose of 200 or higher on oral glucose tolerance testing)
* Glycosuria

PEDIATRIC PILOT STUDY:

INCLUSION CRITERIA:

* Age 6-12 years at enrollment
* Body weight at least 17 kg
* Prepubertal (Tanner stage I breasts in girls, or testicular volumes less than or equal to 3 mL in boys)
* No known active medical conditions

EXCLUSION CRITERIA:

* Current use of prescription or non-prescription medication. Certain exceptions are permitted, including topical medications and vitamins. Other medications may be permitted at the discretion of the investigators.
* Recent (past 2 months) use of drugs that alter glucose metabolism (e.g. metformin), alter gastric pH (e.g. proton pump inhibitors) or gastric emptying (e.g. metoclopramide)
* ALT or AST more than 1.5 times the upper limit of normal
* Known allergy, sensitivity or other contraindication to any study food or drug or its vehicle
* Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to provide assent, and/or the subject s parent/guardian to provide informed consent, or to comply with study procedures
* Abnormal glucose tolerance (fasting blood glucose of 100 mg/dl or higher, or 2-hour blood glucose of 140 or higher on oral glucose tolerance testing)
* Glycosuria

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion change with sucralose | At minute -10,0,10, 20,30,60,90,120
  After a 10-hour fast, subjects will drink a 75-gram oral glucose solution. Samples will be drawn at -10, 0, 10, 20, 30, 60, 90, and 120 minutes.

SECONDARY OUTCOMES:
Change in gastric emptying | At minute -10,0,10, 20,30,60,90,120
  Gastric emptying will be assessed using acetaminophen labeling. For this test, 1450 mg of acetaminophen oral solution (14.5 mL of acetaminophen infant drops, 100 mg/mL) will be mixed with the oral glucose solution or mixed meal. Acetaminophen levels will be measured at the same time points as the primary outcome.
Change in satiety | At minute -10,0,10, 20,30,60,90,120
  Perceived ratings of hunger and satiety will be measured through the use of questionnaires during the OGTT or mixed meal tests. Starting 10 minutes before consumption of the non- nutritive sweetener/placebo, the subject with fill out a Visual Analogue Scale (VAS) which contains questions on hunger and satiety. The VAS will be filled out at -10,0,30, 60, 90, and 120 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Sylvetsky AC, Brown RJ, Blau JE, Walter M, Rother KI. Hormonal responses to non-nutritive sweeteners in water and diet soda. Nutr Metab (Lond). 2016 Oct 21;13:71. doi: 10.1186/s12986-016-0129-3. eCollection 2016. PMID 27777606
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-DK-0163.html